CLINICAL TRIAL: NCT00787280
Title: Diet, Imaging and Energy Balance Trial
Brief Title: Diet, Imaging and Energy Balance Trial (DIET)
Acronym: DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00002610
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
Keywords: obese; overweight; fMRI; Diet
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Ketogenic Diet (LCKD) (Experimental): participants will follow a low carbohydrate ketogenic diet for six weeks
  Interventions: Behavioral: Low Carbohydrate Ketogenic Diet (LCKD)
- Low Fat Diet (LFD) (Experimental): particpants will follow a low fat diet for six weeks
  Interventions: Behavioral: Low Fat Diet (LFD)

INTERVENTIONS:
Behavioral: Low Carbohydrate Ketogenic Diet (LCKD) — participants will follow a low carbohydrate ketogenic diet for six weeks
  Arms: Low Carbohydrate Ketogenic Diet (LCKD)
Behavioral: Low Fat Diet (LFD) — particpants will follow a low fat diet for six weeks
  Arms: Low Fat Diet (LFD)

SUMMARY:
To evaluate whether changes in macronutrient consumption (i.e., switching to a diet low in carbohydrates) can change brain responses to cues depicting foods representing that macronutrient. In addition to answering specific questions regarding the effects of an LCKD, the study will provide general information about relations between brain responses to food cues and a broad arrive of factors including typical diet, food preferences, weight control history and genes.

DETAILED DESCRIPTION:
We propose a parallel arm randomized clinical trial of two diets-a low carbohydrate ketogenic diet (LCKD) and a low fat diet (LFD). Following screening, eligible participants will undergo a six week dietary intervention that will include 7 clinic visits at the Duke Lifestyle Medicine Clinic (Director: Dr. Westman). In addition to the dietary intervention, participants will undergo fMRI scanning on two occasions: once in the week prior to randomization to a diet (Baseline Scan) and after three weeks of following a diet (Post-Diet Scan). During scanning participants will view food cues in order to assess the effects of diet on brain responses to different macronutrient content categories (e.g., High vs. Low Complex Carbohydrate). In addition to scanning measures, we will also record information regarding dietary intake, food preferences, weight, mood, and diet adherence.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18-50 years old, right handed and have a BMI > 27 kg/m². They must be willing to follow either of the two diets.

Exclusion Criteria:

1. weigh over 300lbs.
2. have uncontrolled hypertension (systolic >160mm Hg, diastolic >100mm Hg)
3. have hypotension (systolic <90 mm Hg, diastolic <60 mm Hg)
4. have coronary heart disease, or cardiac rhythm disorder
5. cerebrovascular disease or peripheral vascular disease that requires intensive hyperlipidemic therapy
6. other significant co-morbid illnesses such as liver disease (AST or ALT > 100), kidney disease (serum creatinine > 1.5), cancer, severe emphysema, severe hypertriglyceridemia (TG>500)
7. have diabetes (insulin or diet controlled)
8. have a current psychiatric disease
9. have current alcohol abuse (greater than 12 drinks per week)
10. have current drug abuse (or treatment within the last year)
11. use of psychiatric medications (including antidepressants, anti-anxiety agents, anti-psychotics, "muscle relaxants" or any other drug that influences mood, cognition, or neurotransmitter systems, i.e. dopamine, norepinephrine, acetylcholine, serotonin, GABA, and glutamate)
12. have had or have an eating disorder including anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified, binge eating disorder, or any other form of disordered eating
13. have had any bariatric/weight loss surgery
14. be taking any diet pills (prescription or over the counter)
15. have been on any diet in the last 3 months
16. have any restrictive dietary requirements (including: vegetarians, vegans, or any other dietary restraints)
17. have any food allergies
18. be on an exclusively ethnic diet
19. be females who are pregnant, nursing mothers or likely to become pregnant
20. have any major medical condition that would make participation unsafe (e.g., have pacemaker or other metallic implant (including dental, orthopedic, or IUD), uncomfortable (e.g., chronic pain), confound results (e.g., psychiatric condition)
21. be left handed
22. have glaucoma, color blindness
23. be using experimental or investigational drugs
24. or suffering from claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Compared to individuals in the LFD group, individuals placed on an LCKD will exhibit decreased brain responses to high-carbohydrate food cues. | 1 month

SECONDARY OUTCOMES:
In addition to these questions, we will also examine relations between food consumption acquired from the diaries, genetic factors and brain function. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States